CLINICAL TRIAL: NCT03349515
Title: The Effect of Povidone-iodine Ophthalmic Surgical Prep Solution on Respiration in Children Undergoing Strabismus Surgery With General Anesthesia.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Michelle Rovner, MD, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00067331
Record Dates: First submitted 2017-10-23; First posted 2017-11-21 (Actual); Results first posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Strabismus
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Intervention Model Description: Group A - povidone-iodine ophthalmic solution, or Group B - ophthalmic balanced salt solution. This randomization will be determined using a simple randomization scheme provided by the study's statistician
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A - povidone-iodine ophthalmic solution. (Active Comparator): Group A will receive three drops of povidone-iodine ophthalmic solution in each eye, with the right eye to receive the drops first.
  Interventions: Drug: Provodine-Iodine Solution
- Group B - ophthalmic balanced salt solution. (Active Comparator): Group B will receive three drops in each eye of ophthalmic balanced salt solution, with the right eye to receive the drops first.
  Interventions: Drug: Group B will receive three drops in each eye of ophthalmic balanced salt solution.

INTERVENTIONS:
Drug: Provodine-Iodine Solution — Group A will receive three drops of povidone-iodine ophthalmic solution in each eye, with the right eye to receive the drops first. The eye drops will be administered by the study anesthesiologist. After application of either solution to the eyes of the patient, any change in ventilation can be detected and timed by observation of the capnography (end-tidal carbon dioxide) and direct observation of the chest wall with use of the iPhone stopwatch feature again. The capnograph is a standard monitor of respiration used during the administration of general anesthesia. Data collected at this time will include whether or not there was a change in respiration, what this change in respiration was, if assisted ventilation was required, how long assisted ventilation was required (if applicable), HR, BP, RR, SaO2 , ETCO2, InspSevo, and ExpSevo. This study intervention and data collection will take less than 5 minutes.
  Arms: Group A - povidone-iodine ophthalmic solution.
Drug: Group B will receive three drops in each eye of ophthalmic balanced salt solution. — Group B will receive three drops in each eye of ophthalmic balanced salt solution. The eye drops will be administered by the study anesthesiologist. After application of either solution to the eyes of the patient, any change in ventilation can be detected and timed by observation of the capnography (end-tidal carbon dioxide) and direct observation of the chest wall with use of the iPhone stopwatch feature again. The capnograph is a standard monitor of respiration used during the administration of general anesthesia. Data collected at this time will include whether or not there was a change in respiration, what this change in respiration was, if assisted ventilation was required, how long assisted ventilation was required (if applicable), HR, BP, RR, SaO2 , ETCO2, InspSevo, and ExpSevo. This study intervention and data collection will take less than 5 minutes
  Arms: Group B - ophthalmic balanced salt solution.

SUMMARY:
Determine whether the application of povidone-iodine ophthalmic solution onto the ocular surface causes a change in respiration in children undergoing strabismus surgery with general anesthesia.

Hypothesis: The application of povidone-iodine ophthalmic solution to the ocular surface causes a change in respiration in children during general anesthesia prior to strabismus surgery.

DETAILED DESCRIPTION:
The study is randomized and single blind. One hundred children were randomly assigned to have either povidone-iodine (group A) or balanced salt solution (BSS) (group B) eye drops instilled into their eyes during anesthesia just prior to strabismus surgery. After induction of anesthesia and insertion of an LMA while the patient was at a steady state of anesthesia and spontaneously breathing sevoflurane in oxygen, 3 drops of either povidone-iodine or BSS was instilled into each eye (right eye first). Respiratory rate was determined by measuring the peak-to-peak interval on the capnograph. This is similar to calculating heart rate by measuring the R-R interval on an ECG. HR, BP, SaO2, EtCO2, and expired sevoflurane were measured in each patient. Medical history information collected included history of prior surgeries, co-existing diseases, or apnea. Appropriate statistical analyses were performed for comparisons between the groups with respect to respiratory rate, HR, BP, expired sevoflurane, and co-existing diseases.

ELIGIBILITY:
* Inclusion Criteria

  * Children between the ages of 1 year and 17 years
  * Scheduled for strabismus surgery
  * Anesthesia plan includes inhalational induction with sevoflurane and the use of a laryngeal mask airway (LMA) with spontaneous ventilation, per the attending anesthesiologist.

Exclusion Criteria

* History of an adverse reaction to iodine
* History of any thyroid disease
* Patients who require tracheal intubation, as determined by the attending anesthesiologist; e.g. craniofacial anomalies.
* Patients with a contraindication to sevoflurane, such as malignant hyperthermia or severe left ventricular dysfunction.
* Inability or unwillingness of the subject or legal guardian/ representative to give informed consent.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A - Povidone-iodine Ophthalmic Solution.: Group A will receive three drops of povidone-iodine ophthalmic solution in each eye, with the right eye to receive the drops first.
  The eye drops will be administered by the study anesthesiologist.
Period: Overall Study
Arm/Group | Group A - Povidone-iodine Ophthalmic Solution. | Group B - Ophthalmic Balanced Salt Solution.
Started | 55 | 51
Completed | 50 | 50
Not Completed | 5 | 1
Not completed — Lack of Efficacy | 2 | 0
Not completed — Physician Decision | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A - Povidone-iodine Ophthalmic Solution. | Group B - Ophthalmic Balanced Salt Solution. | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants] — Population: There were 6 patients withdrawn. 5 from Group A and 1 from Group B
  Participants
    <=18 years | 50 | 50 | 100
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: There were 6 participants withdrawn. 5 from Group A and 1 from Group B.
  years | 6.2 (3.9) | 6.4 (3.4) | 6.31 (3.61)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There were 6 participants withdrawn. 5 from Group A and 1 from Group B.
  Participants
    Female | 33 | 27 | 60
    Male | 17 | 23 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: There were 6 participants withdrawn from the study. 5 from Group A and 1 from Group B.
  Participants
    Hispanic or Latino | 3 | 2 | 5
    Not Hispanic or Latino | 47 | 48 | 95
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: There were 6 participants that were withdrawn. 5 from Group A and 1 from Group B.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 8 | 12 | 20
    White | 38 | 35 | 73
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants] — Population: There were 6 participants withdrawn from the study. 5 from Group A and 1 from Group B.
  participants
    United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Breath Duration
Description: The iPhone stopwatch application will be used and its 'lap button' feature to collect the respiration peak intervals (in seconds) for 5 breaths. Specifically, at the patient's peak inspiration (as seen on the capnography), the study member will start the stopwatch and proceed to hit the 'lap' button for the next 5 consecutive inspiration peaks. These data intervals will be recorded on the data sheet after the 5 breaths are over, as the intervals are conveniently stored and numbered below the stopwatch in the app
Time Frame: 5 minutes
Measure: Mean (Standard Error); unit: seconds
Groups:
- Group A - Povidone-iodine Ophthalmic Solution.: Group A will receive three drops of povidone-iodine ophthalmic solution in each eye, with the right eye to receive the drops first. The eye drops will be administered by the study anesthesiologist. After application of either solution to the eyes of the patient, any change in ventilation can be detected and timed by observation of the capnography (end-tidal carbon dioxide) and direct observation of the chest wall with use of the iPhone stopwatch feature again. The capnograph is a standard monitor of respiration used during the administration of general anesthesia. Data collected at this time will include whether or not there was a change in respiration, what this change in respiration was, if assisted ventilation was required, how long assisted ventilation was required (if applicable), HR, BP, RR, SaO2 , ETCO2, InspSevo, and ExpSevo. This study intervention and data collection will take less than 5 minutes.
Arm/Group | Group A - Povidone-iodine Ophthalmic Solution. | Group B - Ophthalmic Balanced Salt Solution.
Number analyzed (Participants) | 50 | 50
seconds
  Breath 1 | 2.14 (0.621) | 2.18 (0.626)
  Breath 2 | 2.26 (0.621) | 2.15 (0.626)
  Breath 3 | 5.02 (0.621) | 2.18 (0.626)
  Breath 4 | 5.65 (0.621) | 2.23 (0.626)
  Breath 5 | 3.08 (0.621) | 2.22 (0.626)
  Breath 6 | 7.47 (0.621) | 2.25 (0.626)
  Breath 7 | 3.22 (0.621) | 2.20 (0.626)
  Breath 8 | 2.49 (0.621) | 2.17 (0.626)
  Breath 9 | 2.69 (0.621) | 2.21 (0.626)
  Breath 10 | 2.49 (0.621) | 2.15 (0.626)
  Breath 11 | 2.35 (0.621) | 2.2 (0.626)
  Breath 12 | 2.15 (0.621) | 2.17 (0.626)
  Breath 13 | 2.12 (0.621) | 2.16 (0.626)
  Breath 14 | 2.14 (0.621) | 2.18 (0.626)
  Breath 15 | 2.09 (0.621) | 2.09 (0.626)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the participants surgery when eye drops were placed. This time frame was less than 30 minutes.
Arm/Group | Group A - Povidone-iodine Ophthalmic Solution. | Group B - Ophthalmic Balanced Salt Solution.
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/51
Other Adverse Events (participants affected / at risk) | 0/55 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT03349515/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT03349515/SAP_001.pdf